CLINICAL TRIAL: NCT03899805
Title: A Phase II Study of Eribulin and Pembrolizumab in Soft Tissue Sarcomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Suzanne George, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-082
Record Dates: First submitted 2019-04-01; First posted 2019-04-02 (Actual); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Sarcoma; Liposarcoma; Leiomyosarcoma; Undifferentiated Pleomorphic Sarcoma
Keywords: Sarcoma
MeSH Terms: conditions — Sarcoma; Liposarcoma; Leiomyosarcoma; Histiocytoma, Malignant Fibrous | interventions — eribulin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Liposarcomas (Experimental): * Participants will receive eribulin intravenously on Day 1 and Day 8
  * Pembrolizumab is administered intravenously Day 1, on a 21-day cycle
  Interventions: Drug: Eribulin; Drug: Pembrolizumab
- Leiomyosarcomas (Experimental): * Participants will receive eribulin intravenously on Day 1 and Day 8
  * Pembrolizumab is administered intravenously Day 1, on a 21-day cycle
  Interventions: Drug: Eribulin; Drug: Pembrolizumab
- Undifferentiated Pleomorphic sarcomas (Experimental): * Participants will receive eribulin intravenously on Day 1 and Day 8
  * Pembrolizumab is administered intravenously Day 1, on a 21-day cycle
  Interventions: Drug: Eribulin; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Eribulin — The ability of chemotherapy to kill cancer cells depends on its ability to halt cell division. Usually, the drugs work by damaging the RNA or DNA that tells the cell how to copy itself in division. If the cells are unable to divide, they die. The faster the cells are dividing, the more likely it is that chemotherapy will kill the cells, causing the tumor to shrink. They also induce cell suicide (self-death or apoptosis).
  Other Names: Halaven
Drug: Pembrolizumab — The drug blocks the PD-1 receptor, preventing binding and activation of PD-L1 and PD-L2. This mechanism causes the activation of T-cell mediated immune responses against tumor cells.
  Other Names: Keytruda

SUMMARY:
This research study is studying a combination of drugs (chemotherapy + Immunotherapy) as a possible treatment for liposarcoma, leiomyosarcoma, or undifferentiated pleomorphic sarcoma that has spread and has not responded to standard treatment.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug, or in the case of this study, combination of drugs, to learn whether the combination of drugs works in treating a specific disease. "Investigational" means that the combination of drugs is being studied.

The primary purpose of this research study is to test the safety and effectiveness of eribulin and pembrolizumab in combination for controlling this cancer

The FDA (the U.S. Food and Drug Administration) has approved eribulin for the treatment of liposarcoma, based on a phase III study that compared eribulin and dacarbazine in the treatment of liposarcoma and leiomyosarcoma. The FDA has not approved pembrolizumab for this specific disease but it has been approved for other uses. A phase II study showed rare responses of liposarcoma and undifferentiated pleomorphic sarcoma to treatment with pembrolizumab. While eribulin in combination with pembrolizumab has not previously been tested in the treatment of liposarcoma, leiomyosarcoma, or undifferentiated pleomorphic sarcoma, other research studies and laboratory experiments and information from those studies suggest that the combination of these drugs may help to stop cancer cells from growing. Chemotherapy treatment with eribulin may increase the response to immunotherapy with pembrolizumab

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed liposarcoma, leiomyosarcoma, or undifferentiated/unclassified pleomorphic sarcoma by a Dana-Farber Cancer Institute or Massachusetts General Hospital pathologist
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, MRI, or calipers by clinical exam. See Section 11 for the evaluation of measurable disease.
* Participants must have received at least one prior line of chemotherapy. No limit on prior lines of therapy.
* Age ≥ 18 years.
* ECOG performance status of 0 or 1 (see Appendix A).
* Participants must have normal organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * Hemoglobin ≥ 8 g/dL within the first 2 weeks prior to the first dose of study drugs, transfusion is allowed.
  * total bilirubin ≤1.5× institutional upper limit of normal (ULN) (except participants with Gilbert Syndrome, who can have total bilirubin <3.0 mg/dL)
  * AST(SGOT)/ALT(SGPT)<2.5 x ULN in a participant with no documented liver metastases; ALT and AST <5.0 x ULN in a participant with documented liver metastases
  * creatinine ≤1.5× ULN OR
  * creatinine clearance ≥50 mL/min/1.73 m2 for participants with creatinine levels above institutional normal (using the Cockcroft-Gault Formula below):
  * Female CrCl = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL
  * Male CrCl = (140 - age in years) x weight in kg 72 x serum creatinine in mg/dL
* Available archival tumor tissue including Formalin-fixed, paraffin embedded (FFPE) or fresh frozen, or be willing to undergo baseline biopsy for tumor tissue correlative biomarker studies.
* The effects of eribulin and pembrolizumab on the developing human fetus are unknown. For this reason, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. A male participant must agree to use a contraception as detailed in Appendix G of this protocol during the treatment period and for at least 20 weeks, corresponding to the time needed to eliminate any study treatments, plus an additional 120 days (a spermatogenesis cycle) after the last dose of study treatment. A female participant is eligible to participate if she is not pregnant (see Appendix G), not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) as defined in Appendix G OR
  * A WOCBP who agrees to follow the contraceptive guidance in Appendix G during the treatment period and for at least 20 weeks plus an additional 30 days (a menstruation cycle) after the last dose of study treatment.
  * WOCBP should use an adequate method to avoid pregnancy for at least 20 weeks plus an additional 30 days after the last dose of investigational drug. Women of childbearing potential must have a negative serum pregnancy test within 72 hours prior to the start of Eribulin and Pembrolizumab. Women must not be breastfeeding. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) do not require contraception. Women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL.
  * Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants who have had standard chemotherapy or radiotherapy within 3 weeks prior to entering the study.
* Participants who have not recovered from adverse events (grade 2 or higher toxicities) due to agents administered, radiotherapy, or surgery more than 3 weeks earlier, with the exception of alopecia.
* Previous treatment with eribulin or any anti-PD-1, PD-L1, or PD-L2 agent, or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
* Participants who are currently participating in or have participated in a study of an investigational agent or have used an investigational device within 3 weeks prior to the first dose of study treatment.
* Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 3 weeks after the last dose of the previous investigational agent.
* Known brain metastases that are untreated, symptomatic or require therapy to control symptoms. Participants with previously diagnosed brain metastases are eligible if they have completed treatment at least 4 weeks prior to registration, are neurologically stable and have not experienced any new neurologic symptoms for the last 4 weeks prior to study entry, and have recovered from the effects of radiotherapy or surgery. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (>10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration. Treatment for brain metastases may have included whole brain radiotherapy, radiosurgery, surgery, or a combination as deemed appropriate by the treating physician.
* Have received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
* Inability to comply with study and/or follow-up procedures.
* History of severe hypersensitivity reaction (≥Grade 3) to any monoclonal antibody.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Eribulin or Pembrolizumab.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations which in the PI's opinion makes it undesirable for the participant to participate in the trial or which would jeopardize compliance with the trial and study requirements.
* Pregnant women (WOCBP who had a positive serum pregnancy test on screening or 72 hours prior to initiation of study protocol) are excluded from this study because the effects of Eribulin and Pembrolizumab on the developing fetus are unknown. There is the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Eribulin and Pembrolizumab, breastfeeding should be discontinued if the mother is treated with Eribulin and Pembrolizumab.
* Because the effects of pembrolizumab on chronic viral infection are not well known, participants should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) (true positive) or known acquired immunodeficiency syndrome (AIDS) or if they have a positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection.
* Participants with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, are excluded. These include but are not limited to participants with a history of immune related neurologic disease such as multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, or myasthenia gravis; participants with a history of systemic autoimmune disease such as SLE, connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, or hepatitis; and participants with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome. These participants should be excluded because of the risk of recurrence or exacerbation of disease. Participants with vitiligo or endocrine deficiencies, including thyroiditis managed with replacement hormones such as physiologic corticosteroids, are eligible. Participants with rheumatoid arthritis or other arthropathies; Sjögren's syndrome; psoriasis controlled with topical medication; or participants with positive serology, such as antinuclear antibodies (ANA) or anti-thyroid antibodies, should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible.
* Participants are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event).
* Participants should be excluded if they have a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses <10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Participants are permitted to use topical, ocular, intraarticular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if <10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
* Participants with a history of pneumonitis or interstitial lung disease.
* History of primary immunodeficiency or solid organ transplantation.
* Participants who have had evidence of active or acute diverticulitis, intra-abdominal abscess, GI obstruction, or fistula or abdominal carcinomatosis (which are known risk factors for bowel perforation) should be evaluated for the potential need for additional treatment before coming on study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne George, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Haddox CL, Nathenson MJ, Mazzola E, Lin JR, Baginska J, Nau A, Weirather JL, Choy E, Marino-Enriquez A, Morgan JA, Cote GM, Merriam P, Wagner AJ, Sorger PK, Santagata S, George S. Phase II Study of Eribulin plus Pembrolizumab in Metastatic Soft-tissue Sarcomas: Clinical Outcomes and Biological Correlates. Clin Cancer Res. 2024 Apr 1;30(7):1281-1292. doi: 10.1158/1078-0432.CCR-23-2250. PMID 38236580

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from June 2019 to February 2021.
Groups:
- Liposarcomas; Leiomyosarcomas; Undifferentiated Pleomorphic Sarcomas: * Participants will receive eribulin intravenously on Day 1 and Day 8
  * Pembrolizumab is administered intravenously Day 1, on a 21-day cycle
  Eribulin: The ability of chemotherapy to kill cancer cells depends on its ability to halt cell division. Usually, the drugs work by damaging the RNA or DNA that tells the cell how to copy itself in division. If the cells are unable to divide, they die. The faster the cells are dividing, the more likely it is that chemotherapy will kill the cells, causing the tumor to shrink. They also induce cell suicide (self-death or apoptosis).
  Pembrolizumab: The drug blocks the PD-1 receptor, preventing binding and activation of PD-L1 and PD-L2. This mechanism causes the activation of T-cell mediated immune responses against tumor cells.
Period: Overall Study
Arm/Group | Liposarcomas | Leiomyosarcomas | Undifferentiated Pleomorphic Sarcomas
Started | 20 | 19 | 18
Completed | 1 | 0 | 1
Not Completed | 19 | 19 | 17
Not completed — Physician Decision | 3 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 2
Not completed — Progressive Disease | 10 | 18 | 12
Not completed — Adverse Event | 3 | 1 | 0
Not completed — Death | 2 | 0 | 0
Not completed — Came off for surgery | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposarcomas | Leiomyosarcomas | Undifferentiated Pleomorphic Sarcomas | Total
Number analyzed (Participants) | 20 | 19 | 18 | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.7 (12.6) | 61.8 (8.8) | 57.1 (11.2) | 60.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 17 | 8 | 33
  Male | 12 | 2 | 10 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 1 | 1
  More than one race | 0 | 1 | 0 | 1
  Other | 1 | 0 | 0 | 1
  White | 18 | 18 | 17 | 53
ECOG Performance Status [Count of Participants; unit: Participants] — PS 0: Fully active, able to carry on all pre-disease performance without restriction, PS 1:Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants
    PS 0 | 11 | 10 | 9 | 30
    PS 1 | 9 | 9 | 9 | 27

OUTCOME MEASURES:

1. Primary Outcome: 12-week Progression Free Survival (PFS)
Description: 12-week PFS was defined as the percent probability estimate at 12 weeks based on the Kaplan-Meier method. PFS is defined as the duration of time from study entry to documented disease progression (PD) requiring removal from the study or death. Participants alive without PD were censored at the earliest of the date of the last disease evaluation or start of new anticancer therapy. Per RECIST 1.1 for target lesions: PD is at least a 20% increase in sum LD, taking as reference the smallest sum on study with at least 5 mm absolute increase. For non-target lesions, progression-free means no new lesions or unequivocal progression on existing non-target lesions or not evaluated.
Time Frame: 12 weeks
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Liposarcomas | Leiomyosarcomas | Undifferentiated Pleomorphic Sarcomas
Number analyzed (Participants) | 20 | 19 | 18
percentage of participants | 69.6 [54.5 to 89.0] | 36.8 [22.5 to 69.4] | 52.6 [36.8 to 75.3]

2. Secondary Outcome: Median Overall Survival (OS)
Description: Overall Survival (OS) based on Kaplan-Meier method is defined as the time from registration to death due to any cause, or censored at date last known alive.
Time Frame: Up to 2 years
Measure: Median (90% Confidence Interval); unit: Weeks
Arm/Group | Liposarcomas | Leiomyosarcomas | Undifferentiated Pleomorphic Sarcomas
Number analyzed (Participants) | 20 | 19 | 18
Weeks | 97.6 [65.4 to NA] — Limited number had events. | 59.1 [38.1 to NA] — Limited number had events. | NA [39.9 to NA] — Limited number had events.

3. Secondary Outcome: Objective Response Rate(ORR)
Description: ORR was defined as the proportion of participants achieving complete response (CR) or partial response (PR) on treatment based on RECIST 1.1 criteria. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Up to 2 years
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Liposarcomas | Leiomyosarcomas | Undifferentiated Pleomorphic Sarcomas
Number analyzed (Participants) | 20 | 19 | 18
proportion of participants | 0.25 [0.104 to 0.456] | 0.47 [0.274 to 0.680] | 0.56 [0.351 to 0.756]

4. Secondary Outcome: Clinical Benefit Response Rate (CBR)
Description: CBR is defined as the proportion of participants who reached stable disease, partical response and complete resposne during treatment based on RECIST 1.1
Time Frame: Up to 2 years
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Liposarcomas | Leiomyosarcomas | Undifferentiated Pleomorphic Sarcomas
Number analyzed (Participants) | 20 | 19 | 18
proportion of participants | 0.75 [0.54 to 0.90] | 0.53 [0.32 to 0.73] | 0.44 [0.24 to 0.66]

ADVERSE EVENTS:
Time Frame: Up to 2 years.
Description: A serious adverse event (SAE) is any adverse event occurring at any dose that, 1) results in death; 2) is life threatening; 3) results in persistent or significant disability/incapacity; 4) results in or prolongs an existing inpatient hospitalization; 5) is a congenital anomaly/birth defect; 6) is a new cancer (that is not a condition of the study); 7) is associated with an overdose; 8) is another important medical event
Arm/Group | Liposarcomas | Leiomyosarcomas | Undifferentiated Pleomorphic Sarcomas
All-Cause Mortality (participants affected / at risk) | 10/20 | 12/19 | 8/18
Serious Adverse Events (participants affected / at risk) | 9/20 | 8/19 | 8/18
Other Adverse Events (participants affected / at risk) | 20/20 | 19/19 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liposarcomas (N=20) | Leiomyosarcomas (N=19) | Undifferentiated Pleomorphic Sarcomas (N=18)
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 0 | 0
Edema limbs (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 0 | 0
Hepatitis viral (Infections and infestations) | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 2 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 3 | 0
Serum amylase increased (Investigations) | 0 | 1 | 0
White blood cell decreased (Investigations) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liposarcomas (N=20) | Leiomyosarcomas (N=19) | Undifferentiated Pleomorphic Sarcomas (N=18)
Anemia (Blood and lymphatic system disorders) | 20 | 19 | 18
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 5 | 1
Eosinophilia (Blood and lymphatic system disorders) | 2 | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 5 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 3 | 1 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 0 | 2
Chest pain - cardiac (Cardiac disorders) | 1 | 1 | 0
Palpitations (Cardiac disorders) | 3 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 4 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 9 | 1 | 9
Ventricular tachycardia (Cardiac disorders) | 0 | 2 | 0
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 | 2 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 1 | 1 | 3
Hyperthyroidism (Endocrine disorders) | 2 | 0 | 2
Hypophysitis (Endocrine disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 3 | 0 | 5
Blurred vision (Eye disorders) | 0 | 1 | 1
Dry eye (Eye disorders) | 0 | 0 | 1
Eye disorders - Other, specify (Eye disorders) | 0 | 1 | 0
Eyelid function disorder (Eye disorders) | 0 | 0 | 2
Optic nerve disorder (Eye disorders) | 1 | 0 | 0
Periorbital edema (Eye disorders) | 3 | 0 | 0
Scleral disorder (Eye disorders) | 0 | 1 | 0
Watering eyes (Eye disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 3 | 1
Belching (Gastrointestinal disorders) | 0 | 1 | 0
Bloating (Gastrointestinal disorders) | 1 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 12 | 5 | 7
Diarrhea (Gastrointestinal disorders) | 13 | 19 | 3
Dry mouth (Gastrointestinal disorders) | 4 | 5 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0 | 5
Flatulence (Gastrointestinal disorders) | 1 | 2 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 4
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 | 2 | 1
Gastroparesis (Gastrointestinal disorders) | 1 | 0 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1
Jejunal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 4 | 7 | 10
Nausea (Gastrointestinal disorders) | 20 | 15 | 15
Oral pain (Gastrointestinal disorders) | 5 | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 3 | 0 | 0
Rectal pain (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 6 | 4 | 2
Chills (General disorders) | 4 | 1 | 3
Edema limbs (General disorders) | 5 | 10 | 6
Fatigue (General disorders) | 20 | 19 | 18
Fever (General disorders) | 5 | 19 | 6
Flu like symptoms (General disorders) | 0 | 4 | 0
Gait disturbance (General disorders) | 1 | 0 | 1
General disorders and administration site conditions - Other, specify (General disorders) | 2 | 4 | 1
Generalized edema (General disorders) | 1 | 0 | 0
Localized edema (General disorders) | 0 | 0 | 3
Non-cardiac chest pain (General disorders) | 0 | 3 | 4
Pain (General disorders) | 9 | 8 | 8
Allergic reaction (Immune system disorders) | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 1
Otitis media (Infections and infestations) | 1 | 0 | 0
Papulopustular rash (Infections and infestations) | 2 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Pleural infection (Infections and infestations) | 0 | 1 | 0
Shingles (Infections and infestations) | 1 | 0 | 1
Skin infection (Infections and infestations) | 1 | 2 | 0
Thrush (Infections and infestations) | 2 | 6 | 2
Tooth infection (Infections and infestations) | 0 | 0 | 2
Upper respiratory infection (Infections and infestations) | 1 | 4 | 1
Urinary tract infection (Infections and infestations) | 2 | 4 | 0
Vulval infection (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 2
Vaccination complication (Injury, poisoning and procedural complications) | 2 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 13 | 17 | 10
Alkaline phosphatase increased (Investigations) | 9 | 14 | 2
Aspartate aminotransferase increased (Investigations) | 15 | 18 | 10
Blood bilirubin increased (Investigations) | 1 | 7 | 0
Blood lactate dehydrogenase increased (Investigations) | 13 | 6 | 18
Cardiac troponin T increased (Investigations) | 1 | 0 | 0
Creatinine increased (Investigations) | 6 | 5 | 3
Electrocardiogram QT corrected interval prolonged (Investigations) | 14 | 0 | 0
Investigations - Other, specify (Investigations) | 0 | 0 | 3
Lipase increased (Investigations) | 18 | 19 | 14
Lymphocyte count decreased (Investigations) | 1 | 0 | 0
Lymphocyte count increased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 20 | 19 | 18
Platelet count decreased (Investigations) | 5 | 11 | 0
Serum amylase increased (Investigations) | 10 | 11 | 6
Thyroid stimulating hormone increased (Investigations) | 2 | 6 | 2
Weight gain (Investigations) | 0 | 1 | 0
Weight loss (Investigations) | 15 | 16 | 10
White blood cell decreased (Investigations) | 20 | 19 | 18
Anorexia (Metabolism and nutrition disorders) | 19 | 17 | 10
Dehydration (Metabolism and nutrition disorders) | 5 | 5 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 20 | 18 | 18
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 | 10 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 6 | 8 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 11 | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 19 | 10 | 7
Hyponatremia (Metabolism and nutrition disorders) | 20 | 17 | 9
Hypophosphatemia (Metabolism and nutrition disorders) | 15 | 5 | 6
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 16 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 6 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 3 | 5
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscle cramp (Musculoskeletal and connective tissue disorders) | 3 | 4 | 9
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 6 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 3 | 3
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Anosmia (Nervous system disorders) | 0 | 0 | 2
Concentration impairment (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 2
Dysgeusia (Nervous system disorders) | 6 | 3 | 8
Headache (Nervous system disorders) | 3 | 7 | 5
Memory impairment (Nervous system disorders) | 0 | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 14 | 8 | 7
Presyncope (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Confusion (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 5 | 8 | 7
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 0 | 3
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 1 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 0 | 1
Urinary urgency (Renal and urinary disorders) | 1 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 0 | 0 | 1
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal pain (Reproductive system and breast disorders) | 0 | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 3 | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 | 6 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 11 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 3
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Nail changes (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 5 | 6
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 | 10 | 7
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 | 11 | 4
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hot flashes (Vascular disorders) | 0 | 2 | 0
Hypertension (Vascular disorders) | 20 | 3 | 10
Hypotension (Vascular disorders) | 1 | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 0
Vascular disorders - Other, specify (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/05/NCT03899805/Prot_SAP_000.pdf